CLINICAL TRIAL: NCT01577823
Title: Utility of Indwelling Catheter in Orthopaedic Patients Receiving Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: RIJPARU2011
Record Dates: First submitted 2011-12-08; First posted 2012-04-16 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Total Joint Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No foley catheter (No Intervention)
- Foley Catheter (Active Comparator)
  Interventions: Device: Foley Catheter

INTERVENTIONS:
Device: Foley Catheter
  Arms: Foley Catheter

SUMMARY:
A study measuring utility of indwelling bladder catheter placement in orthopaedic surgical patients receiving spinal anesthesia. Study will track clinical outcomes, patient satisfaction and cost efficacy. Absence of indwelling bladder catheter may decrease urinary tract infection (UTI) incidence, increase patient satisfaction, and decrease cost burden without increasing postoperative urinary retention (POUR) incidence.

ELIGIBILITY:
Inclusion Criteria:

Elective orthopaedic surgical patients of all ages undergoing lower extremity adult reconstructive surgery with spinal anesthesia will be interviewed.

Exclusion Criteria:

Patients are excluded from the study preoperatively with a history of prostate or urological surgery, renal failure, previous documented POUR, current indwelling catheter, or acute UTI.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States